CLINICAL TRIAL: NCT06394453
Title: Is Feeding During Therapeutic Hypothermia Safe and Can Improve Outcomes in Infants With Hypoxic-ischaemic Encephalopathy: a Randomized Controlled Study.
Brief Title: Is Feeding During Therapeutic Hypothermia Safe and Can Improve Outcomes in Infants With Hypoxic-ischaemic Encephalopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Foundation (Other)
Responsible Party: Principal Investigator, Viktoryia Parfenchyk, Principal Investigator, Physician, Nutricia Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NutriciaFoundation
Record Dates: First submitted 2024-04-20; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Newborn Asphyxia
Keywords: therapeutic hypothermia, hypoxic-ischaemic encephalopathy
MeSH Terms: conditions — Asphyxia Neonatorum; Hypoxia-Ischemia, Brain | interventions — Enteral Nutrition

STUDY DESIGN:
Intervention Model Description: All eligible newborns will be randomized to one of the two groups :
  1. unfed during 72 hours of TH (control group);
  2. fed group, which will start receiving enteral feeding with mother milk or human donor breast milk at 10 ml/kg/day during first day of TH, 20 ml/kg/day during second day and 30 ml/kg/day during third day (experimental group).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Control group will be unfed orally during 72 hours of therapeutic hypothermia. The group will be receiving parenteral nutrition (PN) from day one onwards. Parenteral nutrition will be defined as receiving any type of nutrient solution in any volume through any route of administration (peripheral venous cannula, central venous catheter, or umbilical catheter).
- experimental group (Experimental): Experimental group will start receiving enteral feeding at 10 ml/kg/day during first day of TH, 20 ml/kg/day during second day and 30 ml/kg/day during third day.
  Additionally will be receiving parenteral nutrition (PN) from day one onwards. Parenteral nutrition will be defined as receiving any type of nutrient solution in any volume through any route of administration (peripheral venous cannula, central venous catheter, or umbilical catheter). As the volume of enteral feeding will be increased, the volume of PN will be decreased gradually.
  Interventions: Other: enteral feeding with mother milk or human donor breast milk

INTERVENTIONS:
Other: enteral feeding with mother milk or human donor breast milk — The experimental group will start enteral feeding with mother milk or human donor breast milk if mother milk is not accesible during the first day of therapeutic hypothermia.
  Arms: experimental group

SUMMARY:
Therapeutic hypothermia (TH) is the standard of care for newborns with moderate to severe hypoxic-ischaemic encephalopathy (HIE) born at 35 weeks or more of gestation. Many neonatal units do not use enteral feeding during TH, in fear of increased risk of complications. Withholding enteral feedings during TH lacks supporting evidence. The aim of the study is to determine if enteral feeding during TH in patients with HIE is safe and assess its effects. Investigators will perform multicenter randomized controlled study in level III neonatal intensive care units on infants qualified for TH. Infants will be randomized into 2 groups: (1) unfed during 72 hours of TH; (2) fed group, which will start receive enteral feeding with mother milk or human donor breast milk at 10 ml/kg/day during first day of TH, 20 ml/kg/day during second day, 30 ml/kg/day during third day. The primary outcome will be (1) combined necrotizing enterocolitis or death, (2) length of hospital stay. The secondary outcomes will be (1) time to full enteral feeding, (2) late-onset sepsis, (3) Test of Infant Motor Performance scoring, (4) MRI scoring, (5) MR spectroscopy parameters.

DETAILED DESCRIPTION:
Investigators will perform a multi-centre, randomized, parallel-arm study in level III neonatal intensive care units in southern part of Poland (Małopolska - 3 units and Podkarpacie - 2 units) on infants qualified for TH. A randomization of subjects will be done via computer software (Redcap Randomization Module). Participants will be allocated to an intervention (TH+human milk (HM)) or control (TH) group. In both groups standard therapeutic hypothermia to rectal temperature of 33,5 C will be performed by 72 hours, including during neonatal transport for outborn babies, starting within 6 hours after birth. Investigators will use mother milk or human donor breast milk, if mother milk is not available.

1. Inclusion criteria:

   1. 35 weeks or more gestational age
   2. < 6 hours post birth
   3. Any of the following:

      * Metabolic or mixed acidosis with a pH of ≤7.0 or a base deficit ≥16 mmol/L in an umbilical cord blood sample or any blood obtained within first hour after birth
      * 10-minute Apgar score of ≤5
      * Ongoing resuscitation initiated at birth and continued for ≥10 minutes
   4. Moderate to severe encephalopathy on clinical examination, using a Thompson HIE score ≥ 7
   5. Signed informed consent by parent
2. Exclusion criteria:

   1. Critical general condition;
   2. Aneuploidies (13 th , 18 th , 21 st );
   3. Birth weight <1800 g;
   4. Severe congenital defects with poor prognosis;
   5. Severe mechanical head injuries;
   6. Congenital malformations of digestive system (esophageal atresia, duodenal atresia, gastroschisis, omphalocele, anal atresia).

      All eligible newborns will be randomized to one of the two groups :
      1. unfed during 72 hours of TH (control group);
      2. fed group, which will start receiving enteral feeding with mother milk or human donor breast milk at 10 ml/kg/day during first day of TH, 20 ml/kg/day during second day and 30 ml/kg/day during third day (experimental group).

      Both groups will be receiving parenteral nutrition (PN) from day one onwards. Parenteral nutrition will be defined as receiving any type of nutrient solution in any volume through any route of administration (peripheral venous cannula, central venous catheter, or umbilical catheter). As the volume of enteral feeding will be increased, the volume of PN will be decreased gradually.

      During the feeding process participants will be routinely checked up for the signs of feeding intolerance or NEC. Feeding intolerance (FI) will be defined with the presence of one or more of these criteria: (1) gastric residuals >50% on a single occasion among participants who received nosogastric feeds; (2) bilious/bloody gastric residuals among participants who received nosogastric feeds; (3) abdominal distension (increase in abdominal girth by > 2 cm from baseline); (4) emesis; (5) gross or occult blood in the stool.

      Necrotizing enterocolitis (NEC, Bell stage 2 or 3) will be diagnosed based on the presence of one or more of the clinical signs (bilious gastric aspirate or emesis, abdominal distension, occult or gross blood in stool) and the presence of at least one of the following sonographic findings: (1) pneumatosis intestinalis, (2) portal vein gas and/or (3) pneumoperitoneum.

      The criteria for stopping the trial intervention: (1) any serious adverse events for enteral feeds, mainly including NEC; (2) infant developed severe/unstable condition (e.g. severe pulmonary hypertension), which lead to stop TH and fasting must last for more than 24 hours.

      Primary endpoints: 1) Combined Necrotizing enterocolitis or death. Necrotizing enterocolitis will be defined by the modified Bell's staging criteria (stage II or stage III).

      2) Length of hospital stay assessed as duration of time spent in hospital before discharge, measured in days.

      Secondary endpoints: 1) Time to full enteral feeding, full enteral feeding defined as participants receive all of their prescribed nutrition as milk feeds and do not receive any supplemental parenteral fluids or nutrition 2) Late-onset sepsis, defined as sepsis occurring at or after 72 hours of life 3) Test of Infant Motor Performance scoring 4) MRI scoring, using MRI scoring system by Rutherford et al., classifying the severity of injury in the basal ganglia and thalami (BGT), cortex (CX), white matter (WM) (each on a scale of 0-3) and posterior limb of the internal capsule (PLIC) (scale 0-2), the higher number indicating more severe abnormality. Total injury score (TIS) will be the sum of these regional scores (scale of 0-11).

      5) MR spectroscopy parameters, such as Lac/NAA, Lac/Cr, NAA/Cr, CHO/NAA Primary outcomes are reduction of mortality or NEC stage 2 or 3 and length of hospital stay. Investigators assumed that 50% difference as being a clinically significant. Estimated that 43 children in each group are needed to achieve a significant difference with a power of 90%, along with a two-sided 5% significance level. Given the anticipated dropout rate of 20%, 52 subjects are necessary in each group.

      Participants will be randomly assigned to either control or experimental group with a 1:1 allocation based on a computer-generated randomization (Redcap). Caregivers of the participants will remain unblinded. The researchers and the statistician will be blinded until the end of the study.

      The analyses will be performed after last patient out, after monitoring and cleaning of data gathered from all patients. Analyses will be performed by the investigators and statistician, using the latest version of Medcalc statistics software.

      The flow of participants will be illustrated in a flow diagram according the Consolidation Standard of Reporting Trials (CONSORT).

      The main analysis will be performed according the intention-to-treat (ITT) principle.

      The baseline characteristics of the included patients will be reported per randomization group and shown in a baseline table. Dichotomous variables will be summarised as proportion of patients with the count divided by the total number of evaluated patients. Continuous variables will be summarised as mean with standard deviation in case of normal distribution and as median with interquartile range in case of non-normal distribution. Testing for normality of data distributions will be based on the Shapiro-Wilks test. For continuous variables a footnote will state the number of evaluated patients. Differences in baseline characteristics between study arms will be reported as preferred by the intended journal. Differences between the study arms will be analysed using Fisher test, independent t test or Mann-Whitney test if required by the journal.

      The assessment and analysis of the primary and secondary outcomes will be discussed separately. All continuous data will be checked for normality. For continuous outcomes the mean difference (MD) and for dichotomous outcomes the relative risk (RR) will be calculated. The difference between study groups will be considered statistical significant when the p-value is <0,05, when the 95% CI for RR does not include 1.0 or when 95% CI for MD does not include 0.

ELIGIBILITY:
Inclusion Criteria:

1. 35 weeks or more gestational age
2. < 6 hours post birth
3. Any of the following:

   * Metabolic or mixed acidosis with a pH of ≤7.0 or a base deficit ≥16 mmol/L in an umbilical cord blood sample or any blood obtained within first hour after birth
   * 10-minute Apgar score of ≤5
   * Ongoing resuscitation initiated at birth and continued for ≥10 minutes
4. Moderate to severe encephalopathy on clinical examination, using a Thompson HIE score ≥ 7
5. Signed informed consent by parent

Exclusion Criteria:

1. Critical general condition
2. Aneuploidies (13 th , 18 th , 21 st )
3. Birth weight <1800 g
4. Severe congenital defects with poor prognosis
5. Severe mechanical head injuries
6. Congenital malformations of digestive system (esophageal atresia, duodenal atresia, gastroschisis, omphalocele, anal atresia)

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Combined Necrotizing enterocolitis or death | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, during hospital stay, an average of 8 weeks
  Necrotizing enterocolitis will be defined by the modified Bell's staging criteria (stage II or stage III)
Length of hospital stay | assessed from day of birth until discharge from hospital, an average of 8 weeks

SECONDARY OUTCOMES:
Time to full enteral feeding | assessed from day of birth until discharge from hospital, an average of 8 weeks
  full enteral feeding defined as newborn infants receive all of their prescribed nutrition as milk feeds and do not receive any supplemental parenteral fluids or nutrition
Late-onset sepsis | assessed from day of birth until discharge from hospital, an average of 8 weeks
  defined as sepsis occurring at or after 72 hours of life
Test of Infant Motor Performance scoring | assessed from day of birth until discharge from hospital, an average of 8 weeks
MRI scoring | assessed until the end of the third month of life
  Using MRI scoring system by Rutherford et al., classifying the severity of injury in the basal ganglia and thalami (BGT), cortex (CX), white matter (WM) (each on a scale of 0-3) and posterior limb of the internal capsule (PLIC) (scale 0-2), the higher number indicating more severe abnormality. Total injury score (TIS) will be the sum of these regional scores (scale of 0-11)
MR spectroscopy parameter | assessed until the end of the third month of life
  Lac/NAA.
MR spectroscopy parameter | assessed until the end of the third month of life
  Lac/Cr
MR spectroscopy parameter | assessed until the end of the third month of life
  NAA/Cr
MR spectroscopy parameter | assessed until the end of the third month of life
  CHO/NAA

CONTACTS AND LOCATIONS:
Overall Officials: Viktoryia Parfenchyk, MD, Principal Investigator — Collegium Medicum Jagiellonian University in Cracow
Locations (1):
- University Children's Hospital of Cracow, Neonatal intensive care unit, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No